CLINICAL TRIAL: NCT06177275
Title: The Influence of Vertical Implant Position With Immediate Provisionalization on the Marginal Bone Loss in Thick Versus Thin Phenotype. A Randomized Controlled Clinical Trial.
Brief Title: The Influence of Vertical Implant Position on the Marginal Bone Loss in Thick Versus Thin Phenotype.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mohamed Fouad Shemais, Lecturer in the department of Oral Medicine & Periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHR
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Dental Implant; Vertical Position; Esthetic Zone; Bounded Edentulous Area

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Thin vertical soft tissue biotype, Placement of BLX implants 2 mm sub-crestal (Experimental): In Thin vertical soft tissue biotype, Placement of BLX implants 2 mm sub-crestal in single missing anterior or premolar teeth in the esthetic zone with immediate provisionalization via a straight emergence profile temporary crown on a temporary abutment.
  Interventions: Procedure: Placement of BLX implants 2 mm sub-crestal i
- Thin vertical soft tissue biotype, Placement of BLX implants equicrestal (Active Comparator): In Thin vertical soft tissue biotype, Placement of BLX implants equicrestal in single missing anterior or premolar teeth in the esthetic zone with immediate provisionalization via a straight emergence profile temporary crown on a temporary abutment.
  Interventions: Procedure: Placement of BLX implants equicrestal
- Thick vertical soft tissue biotype, Placement of BLX implants 2 mm sub-crestal (Experimental): In Thick vertical soft tissue biotype, Placement of BLX implants 2 mm sub-crestal in single missing anterior or premolar teeth in the esthetic zone with immediate provisionalization via a straight emergence profile temporary crown on a temporary abutment.
  Interventions: Procedure: Placement of BLX implants 2 mm sub-crestal i
- Thick vertical soft tissue biotype, Placement of BLX implants equicrestal (Active Comparator): In Thick vertical soft tissue biotype, Placement of BLX implants equicrestal in single missing anterior or premolar teeth in the esthetic zone with immediate provisionalization via a straight emergence profile temporary crown on a temporary abutment.
  Interventions: Procedure: Placement of BLX implants equicrestal

INTERVENTIONS:
Procedure: Placement of BLX implants 2 mm sub-crestal i — Placement of BLX implants 2 mm sub-crestal in single missing anterior or premolar teeth in the esthetic zone with immediate provisionalization via a straight emergence profile temporary crown on a temporary abutment.
  Arms: Thick vertical soft tissue biotype, Placement of BLX implants 2 mm sub-crestal; Thin vertical soft tissue biotype, Placement of BLX implants 2 mm sub-crestal
Procedure: Placement of BLX implants equicrestal — Placement of BLX implants equicrestal in single missing anterior or premolar teeth in the esthetic zone with immediate provisionalization via a straight emergence profile temporary crown on a temporary abutment.
  Arms: Thick vertical soft tissue biotype, Placement of BLX implants equicrestal; Thin vertical soft tissue biotype, Placement of BLX implants equicrestal

SUMMARY:
Multiple clinical studies have established high survival rates and tremendous predictability of dental implant treatment (Schiegnitz and Al-Nawas 2018). However, a pleasant esthetic outcome is the patient's primary expectation regarding implants in the esthetic zone (Vermylen et al. 2003)and several esthetic factors have been evaluated to contribute to an esthetic appearance. Among these, the midfacial soft tissue level is considered to be one of the most important factors; Cosyn and co-workers reported that among factors including soft tissue phenotype, the midfacial recession was associated with the position of the implant (Cosyn et al. 2012).

Therefore, subcrestal implant placement has been advocated as it has been associated with the reduction of crestal bone loss in cases with decreased soft tissue thickness. If the vertical soft tissues on the crest of the alveolar ridge are 2 mm or less at the time of implant placement, implants will undergo unavoidable bone resorption by establishing sufficient biologic protection. Another option was proposed by Linkevicius et al, who introduced the subcrestal implant placement as a method to accommodate the problem of thin soft tissues.(Linkevicius et al. 2020).

Limiting the extent of peri-implant bone loss has been recognized for decades to be an important aspect of long-term implant success, and stable peri-implant bone conditions play an important role in maintaining esthetics (Laurell and Lundgren, 2011).

The opinion expressed widely in the scientific literature has been that subcrestal implant placement leads to increased crestal bone resorption. However, clinical studies addressing the implant placement depth in relation to crestal bone have been rare. Data on subcrestal versus crestal placement have mostly come from animal studies. Even fewer data are available regarding the effects of crestal versus subcrestal positioning of platform-switched implants (Cochran et al., 2009).

This study aims to compare the effect of different vertical implant position with immediate provisionalization on marginal bone loss thin and thick vertical tissue biotype.

ELIGIBILITY:
Eligibility criteria:

Inclusion criteria:

* Patients with single missing upper anterior or premolar teeth
* Patients with minimum buccolingual width of 6 mm and mesiodistal width of 6mm
* Patients with healthy systemic conditions.
* Patients older than 18 years.
* Good oral hygiene.
* Accepts one year follow-up period (cooperative patients).
* The patient provides informed consent.
* Adequate Inter-arch space for implant placement.
* Favorable occlusion (no traumatic occlusion).
* Absence of allergy to the prescribed medications.

Exclusion criteria:

* Patients with inadequate bone volume and/ or quality
* Patients with local root remnants
* Patients with inadequate wound healing
* Patients with signs of acute infection related to the area of interest.
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits (Lobbezoo et al., 2006).
* Heavy smokers patients (more than 10 cigarettes per day) (Lambert, Morris and Ochi, 2000).
* Metabolic diseases such as diabetes or hyperthyroidism as well as systemic medications such as chemotherapy or bisphosphonates
* Pregnant or nursing women.
* Uncooperative patients.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Crestal bone loss | 1 year
  Interproximal bone loss will be measured using paralleling cone technique with standardized peri-apical x-ray and bone loss will be measured mesial and distal to the implant by measuring the vertical bone loss from the initial implant position at T3 immediately after implant position and T4 (6 months) and T5 (12 months), ,where interproximal bone loss will be defined as the distance from implant shoulder to the mesial and distal first visible bone-implant contact (fBIC) and (b) bone over the implant platform. One independent and calibrated examiner (A.P.) measured these radiological variables to the nearest 0.1 mm (Pico et al., 2019).

SECONDARY OUTCOMES:
Radiographic horizontal bucco-palatal bone changes | 1 year
  The bucco-palatal width of the alveolar bone will be measured perpendicular to the long axis of the alveolar bone; the 3 measurements will be the at 3 levels implant platform, 2mm and 4 mm . Each measurement will be recorded at different times (at day 0 after finishing the procedure and 12 months post-operatively) (Park et al. 2022).
Radiographic vertical bone changes | 1 year
  Vertical bone height will be measured. Measurement will be taken at highest point of the remaining labial/buccal plate of bone using the implant neck as a reference point. Each measurement will be recorded at different times (at day 0 after finishing the procedure and 12 months post-operatively) and the difference between pre and post-operative measurements will be determined as the gain in labial/buccal vertical bone dimension (Wu et al. 2019
Midfacial recession (MFR): | easured at 6, and 12 months
  Corono-apical distance between the peri-implant soft tissue margin and the cemento-enamel junction (CEJ) of the homologous contralateral tooth. Midfacial recession will be (Zucchelli et al. 2019).
Esthetic evaluation | 1 year
  (The pink esthetic score) 1-14 score
implant survival | 1 year
  A binary outcome, the definition of implant success was based on the clinical and radiographic criteria described by Buser et al. 1990 ;1) absence of clinically detectable implant mobility; 2) absence of pain or any subjective sensation; 3) absence of recurrent peri-implant infection; and 4) absence of persistent radiolucency around the implant after 12 months of loading (Buser, Weber and Lang, 1990)
Emergence Angle | 1 year
  The angle between the tangent line of the restoration at the most coronal point of the buccal mucosa and the implant long axis (Wang et al., 2022).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided